CLINICAL TRIAL: NCT02661009
Title: Human EGFR(Epidermal Growth Factor Receptor) Mutations Quantitative Detection Kit (Real-time Fluorescent PCR Method)
Brief Title: Human EGFR Mutations Quantitative Detection Kit (Real-time Fluorescent PCR Method)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GenoSaber (Industry)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); Sun Yat-sen University (Other); Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EGFR2015-01
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Non Small Cell Lung Cancer; EGFR-TKI Resistant Mutation; EGFR-TKI Sensitizing Mutation
Keywords: NSCLC; EGFR; EGFR-TKI; PCR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Plasma and tissue matching
- predicting clinical efficacy

SUMMARY:
In this clinical trial, investigators select FFPE and plasma samples of non-small cell lung cancer which are used for quantitative detection of four kinds of EGFR(Epidermal Growth Factor Receptor) mutations. By the following two aspects, investigators evaluate the clinical performance of the EGFR quantitative kits.

1. methodology validation: To certify the equivalence between the EGFR quantitative kit and the common used detection methods.
2. analysis of the relationship between the type and proportion of EGFR sensitive mutation and EGFR-TKI benefit.

DETAILED DESCRIPTION:
According to the types of samples and the purpose of the study, the research consists of two groups: plasma and tissue matching group and predicting clinical efficacy group. The samples of the plasma and tissue matching group are the same period plasma and matched FFPE(formalin-fixed paraffin-embedded tissue)samples which will be collected before the first time patients accept any anti-tumor treatment. The samples of predicting clinical efficacy group are FFPE samples which will be collected before the patients receive EGFR-TKI treatment. In addition, the subjects have the complete prognostic follow-up data.

ELIGIBILITY:
Plasma and tissue matching group:

Inclusion Criteria:

* 18~80 years old
* Diagnosis of NSCLC (stage III or IV) which is confirmed by histology or cytology methods.
* Did not receive any anti-tumor treatment.
* Sufficient samples for analysis

Exclusion Criteria:

* Female patients of childbearing potential who are nursing or are pregnant.
* Samples are collected after patients receiving anti-tumor treatment.
* The plasma sample hemolysis.
* Tumor cells are not found in FFPE samples.
* Incomplete information of subjects

predicting clinical efficacy group:

Inclusion Criteria:

* 18~80 years old
* Diagnosis of NSCLC (stage III or IV) which is confirmed by histology or cytology methods.
* At least one measurable focus
* With EGFR-TKI treatment
* Complete follow-up information after EGFR-TKI treatment
* Sufficient samples for analysis

Exclusion Criteria:

* FFPE samples are collected after EGFR-TKI treatment.
* Female patients of childbearing potential who are nursing or are pregnant.
* Tumor cells are not found in FFPE samples.
* Incomplete information of subjects

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non Small Cell Lung Cancer(stage Ⅲ-Ⅳ)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
EGFR mutation detection of FFPE and plasma samples by Human EGFR Mutations Quantitative Detection Kit | 6 months
  Each subject will be collected 3-10 FFPE samples and 3 ml plasma samples.